CLINICAL TRIAL: NCT03791866
Title: The Roles of Th9/IL-9 in the Mechanisms of Early Enteral Nutrition Maintaining Intestinal Mucosal Barrier in Sepsis
Brief Title: The Th9/IL-9 and Early Enteral Nutrition in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, XiangWang, Director, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YKK17102
Record Dates: First submitted 2018-12-21; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Sepsis; Intestinal Mucosal Barrier; Th9 Cells; Enteral Nutrition
MeSH Terms: conditions — Sepsis | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30% target total enteral nutrition (Experimental)
  Interventions: Other: Nutrition
- 60% target total enteral nutrition (Experimental)
  Interventions: Other: Nutrition
- 100% target total enteral nutrition (Active Comparator)
  Interventions: Other: Nutrition

INTERVENTIONS:
Other: Nutrition — Enteral nutrition

SUMMARY:
The investigators aim to evaluate the roles of Th9/IL-9 in the mechanisms of early enteral nutrition (EEN) maintaining intestinal mucosal barrier in sepsis. The results of this study would lay the foundation for revealing the mechanisms of EEN improving immune imbalance of sepsis and provide a new idea to the early treatment of sepsis. In addition, the investigators also aim to evaluate the effects of different proportions of target total enteral nutrition on the prognosis of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of sepsis
2. Within 3 days of sepsis onset before ICU admission
3. No artificial nutrition (enteral or parenteral nutrition) were provided before ICU admission

Exclusion Criteria:

1. Ileus
2. Digestive tract hemorrhage
3. Inflammatory bowel disease
4. Abdominal hypertension (IAP >25mmHg)
5. Cancer or chronic organ dysfunction (e.g., hepatic or renal dysfunction)
6. Malnutrition or immunodeficiency
7. Long-term use of hormones

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
28-d mortality | 28 days

SECONDARY OUTCOMES:
Serum Th9 lymphocyte percentages | 7 days
  Serum Th9 lymphocyte percentages
Concentration of serum IL-9 | 7 days
  Concentration of serum IL-9
Concentration of serum iFABP | 7 days
  Concentration of serum iFABP
Concentration of serum DAO | 7 days
  Concentration of serum DAO

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Kui Sun, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Sun JK, Zhou J, Sun XP, Shen X, Zhu DM, Wang X, Zhou SM, Mu XW. Interleukin-9 promotes intestinal barrier injury of sepsis: a translational research. J Intensive Care. 2021 May 3;9(1):37. doi: 10.1186/s40560-021-00550-y. PMID 33941281